CLINICAL TRIAL: NCT03659630
Title: MyCompass in a Swedish Context - Lessons Learned From the Transfer of an Automated Self-help Intervention Targeting Mental Health Problems
Brief Title: MyCompass in a Swedish Context - an Automated Self-help Intervention Targeting Mental Health Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Clara Hellner Gumpert, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/1268-31/2 + 2016/88
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Mild Depression; Anxiety State; Sleep Disturbance; Stress, Psychological
MeSH Terms: conditions — Anxiety Disorders; Parasomnias; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group receives the MyCompass intervention, an automated self-help intervention for mild to moderate mental ill-health.
  Interventions: Behavioral: MyCompass
- Comparison group (Placebo Comparator): The control group receives a brief email each week, describing the most common mental health issues.
  Interventions: Behavioral: Comparison group

INTERVENTIONS:
Behavioral: MyCompass — Self-help tools to change behaviours in various different domains including sleep deprivation, anxiety and depression.
  Arms: Intervention group
Behavioral: Comparison group — An email containing a brief text on general tips regarding mental health was sent out once a week.
  Arms: Comparison group

SUMMARY:
The study present findings from the implementation of myCompass, a fully automated self-help intervention of Australian origin for mild to moderate anxiety and depression, in a Swedish context. The study also investigates the usage of a specially designed research platform aimed at handling informed consent and online surveys.

ELIGIBILITY:
Inclusion Criteria:

* Swedish resident
* Valid e-mail address
* 18 years old or older
* PHQ-9 score of 5-20
* GAD-7 score of 5-15

Exclusion Criteria:

* suicidal thoughts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 2 weeks
  Self-report measure on depressive symptoms. Nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score, where a higher score indicates more severe depression. Scores of 5, 10, 15, and 20 are taken as the cut-off points for mild, moderate, moderate to severe and severe depression, respectively. For the purpose of this study, participants with a score between 5-20 were included.
Generalised Anxiety Disorder 7-item scale (GAD-7) | 2 weeks
  Self-report measure on anxiety symptoms. Seven items with score 0-21, a higher score indicating more severe anxiety. Cutoffs: Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. For the purpose of this study, participants with a score between 5-15 were included.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nilsson A, Sorman K, Klingvall J, Ovelius E, Lundberg J, Hellner C. MyCompass in a Swedish context - lessons learned from the transfer of a self-guided intervention targeting mental health problems. BMC Psychiatry. 2019 Jan 31;19(1):51. doi: 10.1186/s12888-019-2039-1. PMID 30704424